CLINICAL TRIAL: NCT00812565
Title: Prospective 24-week, Double-blind, Randomised, Placebo-controlled, Multicenter Study Evaluating Safety and Change in Efficacy-related Surrogate Parameters in Patients With Dementia of the Alzheimer's Type Under Treatment With Increasing Dosages of Intravenous Immunoglobulin (Octagam 10%)
Brief Title: Study of Octagam (Intravenous Immunoglobulin [IVIG]) 10% on the Treatment of Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GAM10-04
Record Dates: First submitted 2008-11-10; First posted 2008-12-22 (Estimated); Results first posted 2014-05-05 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-04

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Placebo every 2 weeks (Placebo Comparator): Participants received placebo intravenously every 2 weeks for 24 weeks (total of 12 infusions).
  Interventions: Drug: Placebo
- 0.1 g/kg octagam 10% every 2 weeks (Experimental): Participants received 0.1 g/kg octagam 10% intravenously every 2 weeks for 24 weeks (total of 12 infusions).
  Interventions: Biological: octagam 10%
- 0.25 g/kg octagam 10% every 2 weeks (Experimental): Participants received 0.25 g/kg octagam 10% every 2 weeks for 24 weeks (total of 12 infusions).
  Interventions: Biological: octagam 10%
- 0.4 g/kg octagam 10% every 2 weeks (Experimental): Participants received of 0.4 g/kg octagam 10% every 2 weeks for 24 weeks (total of 12 infusions).
  Interventions: Biological: octagam 10%
- Placebo every 4 weeks (Placebo Comparator): Participants received placebo intravenously every 4 weeks for 20 weeks (total of 6 infusions).
  Interventions: Drug: Placebo
- 0.2 g/kg octagam 10% every 4 weeks (Experimental): Participants received 0.2 g/kg octagam 10% intravenously every 4 weeks for 20 weeks (total of 6 infusions).
  Interventions: Biological: octagam 10%
- 0.5 g/kg octagam 10% every 4 weeks (Experimental): Participants received 0.5 g/kg octagam 10% every 4 weeks for 20 weeks (total of 6 infusions).
  Interventions: Biological: octagam 10%
- 0.8 g/kg octagam 10% every 4 weeks (Experimental): Participants received of 0.8 g/kg octagam 10% every 4 weeks for 20 weeks (total of 6 infusions).
  Interventions: Biological: octagam 10%

INTERVENTIONS:
Drug: Placebo — Commercially available 0.9% isotonic sodium chloride solution.
  Arms: Placebo every 2 weeks; Placebo every 4 weeks
Biological: octagam 10% — octagam 10% was supplied as ready-to-use solutions of human immunoglobulin.
  Other Names: IVIG
  Arms: 0.1 g/kg octagam 10% every 2 weeks; 0.2 g/kg octagam 10% every 4 weeks; 0.25 g/kg octagam 10% every 2 weeks; 0.4 g/kg octagam 10% every 2 weeks; 0.5 g/kg octagam 10% every 4 weeks; 0.8 g/kg octagam 10% every 4 weeks

SUMMARY:
This study evaluated the effect of 6 or 12 infusions of different doses of octagam (intravenous immunoglobulin [IVIG]) 10% on the reduction of amyloid beta peptide (Aβ) in cerebral spinal fluid (CSF) and on the increase of Aβ in blood plasma in patients with mild to moderate Alzheimer's disease.

DETAILED DESCRIPTION:
Participants received 12 infusions of 0.1 g/kg, 0.25 g/kg, or 0.4 g/kg body weight octagam 10% at 2-week intervals (±3 days) or 6 infusions of 0.2 g/kg, 0.5 g/kg, or 0.8 g/kg body weight octagam 10% at 4-week intervals (±5 days). The effect of the infusions on the reduction of Aβ peptide in CSF and the increase of Aβ peptide in blood plasma was evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Probable Alzheimer's Disease (AD) according to the National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria.
* Age of 50 to 85.
* Mini-mental State Examination (MMSE) score of 16 to 26.
* Sufficient language skills for testing.
* Sufficient vision and hearing for testing.
* Modified Hachinski-Rosen Score < 5.
* Magnetic resonance imaging (MRI) of the head consistent with the diagnosis of AD.
* Caregiver available with contact at least 4 days per week for greater than 1 hour.
* Outpatient status or assisted living.
* Post-menopause (women) as evidenced by lack of menstruation for at least 12 consecutive months or by having bilateral oophorectomy.
* Stable doses of approved AD medication(s) for at least 3 months prior to screening (eg, acetylcholine esterase (AChE) inhibitors, memantine).
* Normal vital signs or clinically insignificant, if outside normal limits.
* Laboratory findings within normal limits or clinically insignificant, if outside normal limits.
* Normal electrocardiogram (ECG) or clinically not significant, if outside normal limits.

Exclusion Criteria:

* Other causes of dementia (eg, vascular dementia, Lewy-body dementia, fronto-temporal dementia, Creutzfeldt-Jacob disease, Huntington's disease, Parkinson's disease).
* History of or present significant other diseases of the central nervous system (eg, brain tumor, normal pressure hydrocephalus, Parkinson's Disease, stroke, severe brain trauma, brain surgery, epilepsy, encephalitis).
* Geriatric depression scale score > 7 (short form with scale from 0 to 15).
* Present significant psychiatric disorder (eg, major depression).
* History of psychosis or hallucinations.
* Mental retardation.
* Unstable medical disease in the opinion of the investigator.
* Insulin dependent diabetes mellitus.
* Acute infectious disease.
* Vitamin B12 deficiency unless on stable replacement therapy for at least 3 months is acceptable.
* Unstable thyroid dysfunction.
* Uncontrolled hypertension.
* Severe liver or kidney disease.
* Major surgery within 3 months prior to screening.
* Prohibited medications: Antiepileptic drugs, antipsychotics (but allowed for treatment of acute episodes), antiparkinson agents, anticholinergic drugs, selegiline, monoamine oxidase inhibitors (MAOI), tricyclics, immunosuppressive medications, anti-histamines (unless on a stable dose for at least 3 months or used for treatment of acute episodes), benzodiazepines (but allowed for treatment of acute episodes), and lithium.
* Antidepressants are permitted, if on a stable dose for at least 3 months and without significant anticholinergic side-effects.
* Peripheral venous conditions which impair establishing regular venous access for infusions.
* Potential reasons that patient may become non-evaluable during the study (eg, planned moving into a nursing home, but assisted living is acceptable).
* Peripheral venous conditions, which impair establishing regular venous access for infusions.
* Known IgA deficiency with antibodies to IgA.
* History of hypersensitivity to blood or plasma derived products, or any component of octagam 10%, such as maltose.
* Medical conditions which interfere with protein catabolism (eg, nephrotic syndrome).
* Known blood hyperviscosity or other hypercoagulable states.
* Deep vein thrombosis within preceding 4 years.
* Symptomatic stroke.
* Transient ischemic attack (TIA) within preceding 2 years.
* Participation in another drug trial within the previous 3 months before screening.
* Participation in immunological treatment studies of AD other than with intravenous immunoglobulin (IGIV) within the previous 6 months before screening.
* IGIV use in the previous 6 months.
* Live viral vaccination within the last month before study entry.
* Not eligible for lumbar puncture (anticoagulant therapy, coagulation disorders, severe spinal alterations).
* Patients with a past or present history of drug abuse or alcohol abuse within the preceding 5 years.
* Patients with any condition that would make the patient, in the opinion of the Investigator, unsuitable for the study.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2009-02; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Frenzel, MD, Study Director — Octapharma Pharmazeutika Produktionsges.m.b.H., Vienna, Austria
Locations (1):
- Octapharma USA, Hoboken, New Jersey, United States

REFERENCES:
- [Derived] Dodel R, Rominger A, Bartenstein P, Barkhof F, Blennow K, Forster S, Winter Y, Bach JP, Popp J, Alferink J, Wiltfang J, Buerger K, Otto M, Antuono P, Jacoby M, Richter R, Stevens J, Melamed I, Goldstein J, Haag S, Wietek S, Farlow M, Jessen F. Intravenous immunoglobulin for treatment of mild-to-moderate Alzheimer's disease: a phase 2, randomised, double-blind, placebo-controlled, dose-finding trial. Lancet Neurol. 2013 Mar;12(3):233-43. doi: 10.1016/S1474-4422(13)70014-0. Epub 2013 Jan 31. PMID 23375965

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was enrolled February 2, 2009. The last patient study visit was September 21, 2010. Patients were enrolled in this study from a variety of settings including private practice clinics and hospitals. There were 12 study sites, 5 in Germany and 7 in the United States.
Pre-assignment Details: Qualified patients meeting all inclusion exclusion criteria and providing informed consent were enrolled into the trial.
Period: Overall Study
Arm/Group | Placebo Every 2 Weeks | 0.1 g/kg Octagam 10% Every 2 Weeks | 0.25 g/kg Octagam 10% Every 2 Weeks | 0.4 g/kg Octagam 10% Every 2 Weeks | Placebo Every 4 Weeks | 0.2 g/kg Octagam 10% Every 4 Weeks | 0.5 g/kg Octagam 10% Every 4 Weeks | 0.8 g/kg Octagam 10% Every 4 Weeks
Started | 8 | 7 | 7 | 7 | 7 | 7 | 8 | 7
Completed | 5 | 6 | 7 | 5 | 6 | 6 | 8 | 6
Not Completed | 3 | 1 | 0 | 2 | 1 | 1 | 0 | 1
Not completed — Did Not Receive Study Medication | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Not completed — Did Not Come to Study Visit | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal of Consent | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Reason Not Specified | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set: All randomized patients who received at least 1 infusion of the study medication and had at least 1 post-baseline efficacy assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Every 2 Weeks | 0.1 g/kg Octagam 10% Every 2 Weeks | 0.25 g/kg Octagam 10% Every 2 Weeks | 0.4 g/kg Octagam 10% Every 2 Weeks | Placebo Every 4 Weeks | 0.2 g/kg Octagam 10% Every 4 Weeks | 0.5 g/kg Octagam 10% Every 4 Weeks | 0.8 g/kg Octagam 10% Every 4 Weeks | Total
Number analyzed (Participants) | 7 | 6 | 7 | 7 | 7 | 6 | 8 | 7 | 55
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.6 (9.2) | 66.8 (5.5) | 68.3 (4.2) | 72.9 (5.0) | 71.4 (11.8) | 74.8 (5.5) | 65.9 (10.2) | 68.4 (8.6) | 70.0 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 3 | 3 | 5 | 2 | 3 | 3 | 24
  Male | 3 | 5 | 4 | 4 | 2 | 4 | 5 | 4 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change in the Area Under the Curve of Plasma Aβ1-40 in the 2 or 4 Weeks After the Last Treatment Infusion From the Trough Level Prior to the Last Treatment Infusion
Description: For participants who received infusions every 2 weeks, plasma samples were collected at the trough level at Week 22 and on Days 1, 4, 7, and 14 after Week 22. For participants who received infusions every 4 weeks, plasma samples were collected at the trough level at Week 20 and on Days 1, 4, 7, 14, 21, and 28 after Week 20. Samples for determining Aβ1-40 in blood plasma were processed at a central laboratory using a commercially available kit from Innogenetics NV (INNO-BIA plasma Aβ forms; Gent, Belgium).
Time Frame: Week 22 to Week 24 for participants who received infusions every 2 weeks and Week 20 to Week 24 participants who received infusions every 4 weeks
Population: Full analysis set: All randomized participants who received at least 1 infusion of the study medication and had at least 1 post-baseline efficacy assessment. Only participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: (pg/mL)*days
Arm/Group | Placebo Every 2 Weeks | 0.1 g/kg Octagam 10% Every 2 Weeks | 0.25 g/kg Octagam 10% Every 2 Weeks | 0.4 g/kg Octagam 10% Every 2 Weeks | Placebo Every 4 Weeks | 0.2 g/kg Octagam 10% Every 4 Weeks | 0.5 g/kg Octagam 10% Every 4 Weeks | 0.8 g/kg Octagam 10% Every 4 Weeks
Number analyzed (Participants) | 5 | 6 | 7 | 5 | 6 | 6 | 8 | 6
(pg/mL)*days | 161.20 (93.90) | -245.67 (747.58) | -122.50 (478.31) | -39.10 (172.72) | 510.92 (2395.80) | -83.67 (957.69) | -755.38 (2232.87) | -262.92 (671.37)

2. Secondary Outcome: Change in Plasma Concentration of Aβ1-40 and Aβ1-42 From Baseline to the End of the Study (Week 24)
Description: Samples for determining Aβ1-40 and Aβ1-42 in blood plasma were processed at a central laboratory using a commercially available kit from Innogenetics NV (INNO-BIA plasma Aβ forms; Gent, Belgium).
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo Every 2 Weeks | 0.1 g/kg Octagam 10% Every 2 Weeks | 0.25 g/kg Octagam 10% Every 2 Weeks | 0.4 g/kg Octagam 10% Every 2 Weeks | Placebo Every 4 Weeks | 0.2 g/kg Octagam 10% Every 4 Weeks | 0.5 g/kg Octagam 10% Every 4 Weeks | 0.8 g/kg Octagam 10% Every 4 Weeks
Number analyzed (Participants) | 7 | 6 | 6 | 6 | 6 | 6 | 7 | 6
pg/mL
  Aβ1-40 | 27.1 (40.2) | 5.5 (64.5) | -0.3 (22.1) | -6.5 (61.4) | -6.0 (23.8) | -20.3 (29.2) | 15.7 (29.7) | -30.5 (42.3)
  Aβ1-42 | 4.1 (3.8) | -2.3 (7.8) | -4.5 (6.3) | -2.7 (7.6) | -2.0 (4.8) | -3.5 (5.8) | -0.1 (4.4) | -7.0 (6.2)

3. Secondary Outcome: Change in Plasma Concentration of Anti-Aβ Autoantibodies From Baseline to the End of the Study (Week 24)
Description: Samples for determining anti-Aβ autoantibodies in blood plasma were processed at a central laboratory using a commercially available kit from DRG Instruments GmbH, (EIA-5099; Marburg, Germany) using methods established at the Department of Neurology, Philipps-University, Marburg, Germany (Professor Dr. med. Richard Dodel). The kit includes 6 standard concentrations of anti-Aβ antibody against which the results of the assay are compared. The standards contain 1, 5, 15, 30, 60, and 120 Relative Units (RTU) which contain 0.03, 0.17, 0.5, 1, 2, and 4 mg IgG/mL, respectively.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: RTU
Arm/Group | Placebo Every 2 Weeks | 0.1 g/kg Octagam 10% Every 2 Weeks | 0.25 g/kg Octagam 10% Every 2 Weeks | 0.4 g/kg Octagam 10% Every 2 Weeks | Placebo Every 4 Weeks | 0.2 g/kg Octagam 10% Every 4 Weeks | 0.5 g/kg Octagam 10% Every 4 Weeks | 0.8 g/kg Octagam 10% Every 4 Weeks
Number analyzed (Participants) | 7 | 6 | 7 | 6 | 6 | 6 | 8 | 6
RTU | 109.7 (284.8) | 74.3 (35.0) | 163.9 (136.6) | 310.2 (193.0) | -56.3 (58.3) | 96.7 (133.7) | 256.6 (214.1) | 501.3 (514.6)

4. Secondary Outcome: Change in the Area Under the Curve of Plasma Aβ1-42 in the 2 or 4 Weeks After the Last Treatment Infusion From the Trough Level Prior to the Last Treatment Infusion
Description: For participants who received infusions every 2 weeks, plasma samples were collected at the trough level at Week 22 and on Days 1, 4, 7, and 14 after Week 22. For participants who received infusions every 4 weeks, plasma samples were collected at the trough level at Week 20 and on Days 1, 4, 7, 14, 21, and 28 after Week 20. Samples for determining Aβ1-42 in blood plasma were processed at a central laboratory using a commercially available kit from Innogenetics NV (INNO-BIA plasma Aβ forms; Gent, Belgium).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: (pg/mL)*days
Arm/Group | Placebo Every 2 Weeks | 0.1 g/kg Octagam 10% Every 2 Weeks | 0.25 g/kg Octagam 10% Every 2 Weeks | 0.4 g/kg Octagam 10% Every 2 Weeks | Placebo Every 4 Weeks | 0.2 g/kg Octagam 10% Every 4 Weeks | 0.5 g/kg Octagam 10% Every 4 Weeks | 0.8 g/kg Octagam 10% Every 4 Weeks
Number analyzed (Participants) | 5 | 6 | 7 | 5 | 6 | 6 | 8 | 6
(pg/mL)*days | 40.70 (48.54) | -8.92 (61.71) | -53.94 (61.59) | -17.00 (23.67) | 50.13 (233.87) | -8.98 (213.29) | -191.58 (456.83) | -64.75 (148.29)

5. Secondary Outcome: Change in the Area Under the Curve of Plasma Anti-Aβ Autoantibodies in the 2 or 4 Weeks After the Last Treatment Infusion From the Trough Level Prior to the Last Treatment Infusion
Description: For participants who received infusions every 2 weeks, plasma samples were collected at the trough level at Week 22 and on Days 1, 4, 7, and 14 after Week 22. For participants who received infusions every 4 weeks, plasma samples were collected at the trough level at Week 20 and on Days 1, 4, 7, 14, 21, and 28 after Week 20. Samples for determining anti-Aβ autoantibodies in blood plasma were processed at a central laboratory using a commercially available kit from DRG Instruments GmbH, (EIA-5099; Marburg, Germany) using methods established at the Department of Neurology, Philipps-University, Marburg, Germany (Professor Dr. med. Richard Dodel). The kit includes 6 standard concentrations of anti-Aβ antibody against which the results of the assay are compared. The standards contain 1, 5, 15, 30, 60, and 120 Relative Units (RTU) which contain 0.03, 0.17, 0.5, 1, 2, and 4 mg IgG/mL, respectively.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: RTU*days
Arm/Group | Placebo Every 2 Weeks | 0.1 g/kg Octagam 10% Every 2 Weeks | 0.25 g/kg Octagam 10% Every 2 Weeks | 0.4 g/kg Octagam 10% Every 2 Weeks | Placebo Every 4 Weeks | 0.2 g/kg Octagam 10% Every 4 Weeks | 0.5 g/kg Octagam 10% Every 4 Weeks | 0.8 g/kg Octagam 10% Every 4 Weeks
Number analyzed (Participants) | 5 | 6 | 7 | 5 | 6 | 6 | 8 | 6
RTU*days | 2829.0 (3957.9) | 358.3 (435.8) | 1862.5 (1470.9) | 2189.6 (2289.3) | 196.6 (1023.0) | 849.4 (2313.6) | 6350.8 (3464.9) | 8494.9 (2292.4)

6. Secondary Outcome: Change From Baseline in Aβ1-40 and Aβ1-42 in Cerebral Spinal Fluid 24-48 Hours After the Last Infusion
Description: Samples for determining Aβ1-40 and Aβ1-42 in cerebral spinal fluid were processed at a central laboratory using a commercially available kit from Meso Scale Discovery (MSD 96-Well Multi-Spot Human/Rodent (4G8) Abeta Triplex Ultra-Sensitive Assay; Rockville, MD, USA).
Time Frame: Baseline to Week 23 Day 2 for participants who received infusions every 2 weeks and Baseline to Week 21 Day 2 for participants who received infusions every 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo Every 2 Weeks | 0.1 g/kg Octagam 10% Every 2 Weeks | 0.25 g/kg Octagam 10% Every 2 Weeks | 0.4 g/kg Octagam 10% Every 2 Weeks | Placebo Every 4 Weeks | 0.2 g/kg Octagam 10% Every 4 Weeks | 0.5 g/kg Octagam 10% Every 4 Weeks | 0.8 g/kg Octagam 10% Every 4 Weeks
Number analyzed (Participants) | 5 | 6 | 7 | 5 | 6 | 6 | 8 | 6
pg/mL
  Aβ1-40 | 939.4 (1670.8) | 266.7 (996.0) | 10.6 (1104.0) | -147.0 (1067.9) | 42.0 (874.0) | 561.7 (1195.5) | 403.9 (588.1) | 642.2 (1171.3)
  Aβ1-42 | 32.4 (67.0) | -8.7 (38.2) | 9.7 (54.7) | 4.0 (40.3) | -5.2 (36.3) | 18.8 (40.3) | 10.5 (40.9) | 24.7 (43.2)

7. Secondary Outcome: Change From Baseline in Anti-Aβ Autoantibodies in Cerebral Spinal Fluid 24-48 Hours After the Last Infusion
Description: as for outcome 3
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: RTU
Arm/Group | Placebo Every 2 Weeks | 0.1 g/kg Octagam 10% Every 2 Weeks | 0.25 g/kg Octagam 10% Every 2 Weeks | 0.4 g/kg Octagam 10% Every 2 Weeks | Placebo Every 4 Weeks | 0.2 g/kg Octagam 10% Every 4 Weeks | 0.5 g/kg Octagam 10% Every 4 Weeks | 0.8 g/kg Octagam 10% Every 4 Weeks
Number analyzed (Participants) | 5 | 6 | 7 | 5 | 6 | 6 | 8 | 6
RTU | 0.38 (3.72) | 0.22 (1.83) | 1.86 (1.93) | -0.78 (1.64) | 0.15 (0.29) | 0.40 (1.43) | 1.12 (1.48) | 0.74 (2.32)

8. Secondary Outcome: Change From Baseline in Tau and Phosphorylated Tau in Cerebral Spinal Fluid 24-48 Hours After the Last Infusion
Description: Samples for determining tau and phosphorylated tau in cerebral spinal fluid were processed at a central laboratory using commercially available kits from Innogenetics NV (INNOTEST® hTau Ag, INNOTEST PHOSPHO-TAU (181P); Gent, Belgium). To measure phosphorylated tau, tau phosphorylated at threonine 181 (pTau181) was determined.
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo Every 2 Weeks | 0.1 g/kg Octagam 10% Every 2 Weeks | 0.25 g/kg Octagam 10% Every 2 Weeks | 0.4 g/kg Octagam 10% Every 2 Weeks | Placebo Every 4 Weeks | 0.2 g/kg Octagam 10% Every 4 Weeks | 0.5 g/kg Octagam 10% Every 4 Weeks | 0.8 g/kg Octagam 10% Every 4 Weeks
Number analyzed (Participants) | 5 | 6 | 7 | 5 | 6 | 6 | 8 | 6
pg/mL
  Tau | 17.4 (38.6) | 209.3 (416.0) | -3.4 (35.6) | -7.8 (51.3) | -33.2 (69.7) | -141.8 (419.5) | 1.3 (86.7) | 131.3 (301.0)
  Phosphorylated tau | 0.60 (7.50) | -3.17 (14.66) | 0.43 (3.60) | 2.60 (4.98) | -1.33 (10.05) | 3.33 (21.23) | -2.50 (8.62) | 10.17 (19.28)

9. Secondary Outcome: Change From Baseline in the Mini Mental Status Examination (MMSE) Score at Week 12 and Week 24
Description: The MMSE test contains 30 questions that assess 8 cognitive domains (orientation to time, orientation to place, registration, attention and calculation, recall, language, repetition, and complex commands). The test is administered by a neuropsychologist, psychometrician, or certified study coordinator. The total score ranges from 0 (severe impairment) to 30 (no impairment), with a higher score indicating a better mental status. A positive change score indicates improvement.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo Every 2 Weeks | 0.1 g/kg Octagam 10% Every 2 Weeks | 0.25 g/kg Octagam 10% Every 2 Weeks | 0.4 g/kg Octagam 10% Every 2 Weeks | Placebo Every 4 Weeks | 0.2 g/kg Octagam 10% Every 4 Weeks | 0.5 g/kg Octagam 10% Every 4 Weeks | 0.8 g/kg Octagam 10% Every 4 Weeks
Number analyzed (Participants) | 7 | 6 | 7 | 6 | 7 | 6 | 8 | 7
Units on a scale
  Week 12 (n=6,6,7,5,7,6,8,7) | 1.5 (2.1) | -2.3 (3.5) | -0.6 (3.0) | -2.0 (3.1) | -0.7 (3.0) | -1.2 (2.3) | -0.3 (2.8) | -0.9 (2.4)
  Week 24 (n=7,6,7,6,6,6,8,6) | -0.7 (3.0) | -2.2 (4.4) | 0.6 (2.5) | -1.7 (2.3) | -1.8 (5.5) | -3.2 (3.3) | -1.8 (1.8) | -1.5 (3.1)

10. Secondary Outcome: Change From Baseline in the Alzheimer's Disease Assessment Scale, Cognitive Part (ADAS Cog) Score at Week 12 and Week 24
Description: The ADAS cog consists of 11 items that assess cognitive areas that are often impaired in Alzheimer's disease, specifically learning (word list), naming (objects), following commands (1 to 5 elements), ideational praxis (mail a letter), constructional praxis (copy 4 figures), orientation (person, time and place), recognition memory (from a second word list), and remembering test instructions (from the recognition subtest). The test includes 3 additional subjective scales that assess spoken language ability, word finding difficulty, and comprehension. The test is administered by a neuropsychologist, psychometrician, or certified study coordinator. The total score ranges from 0 to 70 with a higher score indicating greater cognitive impairment. A negative change score indicates improvement.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo Every 2 Weeks | 0.1 g/kg Octagam 10% Every 2 Weeks | 0.25 g/kg Octagam 10% Every 2 Weeks | 0.4 g/kg Octagam 10% Every 2 Weeks | Placebo Every 4 Weeks | 0.2 g/kg Octagam 10% Every 4 Weeks | 0.5 g/kg Octagam 10% Every 4 Weeks | 0.8 g/kg Octagam 10% Every 4 Weeks
Number analyzed (Participants) | 7 | 6 | 7 | 6 | 7 | 6 | 8 | 7
Units on a scale
  Week 12 (n=6,6,7,5,7,6,8,7) | 1.11 (4.10) | 0.94 (7.27) | -0.86 (4.75) | -0.07 (4.43) | 1.52 (5.67) | 3.67 (3.85) | 1.54 (6.63) | 2.28 (5.06)
  Week 24 (n=7,6,7,6,5,6,8,6) | -0.62 (3.86) | 2.06 (3.32) | -2.14 (4.41) | 3.67 (4.85) | 0.93 (3.29) | 4.17 (4.85) | 3.00 (9.37) | 1.89 (8.71)

11. Secondary Outcome: Change From Baseline in the Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADAS-ADL) Score at Week 12 and Week 24
Description: The ADAS-ADL consists of 23 questions that measure the ability of a person to perform basic activities of daily living, such as eating, walking, bathing, grooming, and dressing. The test is administered by a neuropsychologist, psychometrician, or certified study coordinator. The total score ranges from 0 to 78 with a lower score indicating more impaired ability. A positive change score indicates improvement.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo Every 2 Weeks | 0.1 g/kg Octagam 10% Every 2 Weeks | 0.25 g/kg Octagam 10% Every 2 Weeks | 0.4 g/kg Octagam 10% Every 2 Weeks | Placebo Every 4 Weeks | 0.2 g/kg Octagam 10% Every 4 Weeks | 0.5 g/kg Octagam 10% Every 4 Weeks | 0.8 g/kg Octagam 10% Every 4 Weeks
Number analyzed (Participants) | 7 | 6 | 7 | 6 | 7 | 6 | 8 | 7
Units on a scale
  Week 12 (n=6,6,7,5,7,6,8,7) | 6.7 (4.0) | 0.0 (5.4) | 1.7 (2.8) | -1.2 (3.5) | -0.6 (8.5) | -8.2 (11.8) | 1.8 (5.0) | -1.9 (3.5)
  Week 24 (n=7,6,7,6,5,6,8,6) | 1.9 (5.0) | -1.5 (5.2) | -4.1 (6.6) | -6.5 (9.7) | -1.8 (6.0) | -4.3 (14.4) | 1.5 (8.2) | -1.2 (3.3)

12. Secondary Outcome: Change From Baseline in the Clinical Dementia Ratio, Sum of Boxes (CDR-SOB) Score at Week 12 and Week 24
Description: A semi-structured interview was conducted by a physician, neuropsychologist, psychometrician, or certified study coordinator with the patient and a caregiver. Based on the results of the interview, the patient was rated on 6 domains of cognition and function: Memory, orientation, judgment/problem solving, community activities, home and hobbies, and personal care. Each domain is rated from 0 = no dementia; 0.5 = questionable dementia, mild cognitive impairment; 1 = mild dementia; 2 = moderate dementia; 3 = severe dementia. The total score ranges from 0 to 18 with a higher score indicating more dementia. A negative change score indicates improvement.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo Every 2 Weeks | 0.1 g/kg Octagam 10% Every 2 Weeks | 0.25 g/kg Octagam 10% Every 2 Weeks | 0.4 g/kg Octagam 10% Every 2 Weeks | Placebo Every 4 Weeks | 0.2 g/kg Octagam 10% Every 4 Weeks | 0.5 g/kg Octagam 10% Every 4 Weeks | 0.8 g/kg Octagam 10% Every 4 Weeks
Number analyzed (Participants) | 7 | 6 | 7 | 6 | 7 | 6 | 8 | 7
Units on a scale
  Week 12 (n=6,6,7,5,7,6,8,7) | -0.67 (1.08) | -0.25 (0.76) | 0.21 (0.86) | 0.60 (0.89) | -0.36 (1.38) | 0.42 (1.36) | 0.50 (1.46) | 0.21 (1.52)
  Week 24 (n=7,6,7,6,5,6,8,6) | -0.57 (1.57) | 0.92 (2.15) | 0.14 (1.28) | 1.25 (1.97) | -1.50 (2.55) | 0.83 (1.44) | 0.44 (1.92) | 0.58 (1.66)

13. Secondary Outcome: Change From Screening in Whole Brain and Hippocampal Volume at Week 12 and Week 24
Description: The volume of the whole brain and of the left and right hippocampus was measured using high-resolution structural coronal 3D heavily T1-weighted gradient-echo sequence magnetic resonance imaging. All evaluations were done centrally by Professor Frederik Barkhof at the Image Analysis Centre, VU Medical Center, Amsterdam, Netherlands. A negative change score indicates loss of brain volume.
Time Frame: Screening to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Placebo Every 2 Weeks | 0.1 g/kg Octagam 10% Every 2 Weeks | 0.25 g/kg Octagam 10% Every 2 Weeks | 0.4 g/kg Octagam 10% Every 2 Weeks | Placebo Every 4 Weeks | 0.2 g/kg Octagam 10% Every 4 Weeks | 0.5 g/kg Octagam 10% Every 4 Weeks | 0.8 g/kg Octagam 10% Every 4 Weeks
Number analyzed (Participants) | 5 | 6 | 7 | 5 | 7 | 6 | 8 | 7
cm^3
  Whole brain - Week 12 (n=5,5,7,4,7,6,7,7) | -0.112 (0.738) | -0.548 (1.001) | -0.709 (1.026) | -1.833 (2.001) | 0.533 (0.481) | -0.528 (1.873) | -0.177 (1.219) | -1.109 (0.731)
  Left hippocampus - Week 12 (n=5,6,7,5,7,6,7,7) | -4.3 (2.7) | -3.1 (3.1) | -2.4 (1.7) | -1.8 (4.2) | -2.8 (2.6) | -2.8 (3.9) | -4.8 (5.0) | -2.2 (3.7)
  Right hippocampus - Week 12 (n=5,6,7,5,7,6,7,7) | -3.8 (2.7) | -2.6 (3.8) | -3.6 (2.6) | -3.0 (2.4) | -4.8 (4.2) | -1.8 (1.6) | -1.5 (3.6) | -4.9 (3.2)
  Whole brain - Week 24 (n=4,5,6,5,4,6,8,6) | -1.403 (0.978) | -1.978 (0.798) | -1.488 (0.726) | -1.390 (1.678) | -0.875 (0.780) | -1.363 (1.752) | -1.096 (1.004) | -1.583 (1.070)
  Left hippocampus - Week 24 (n=4,6,6,5,5,6,8,6) | -7.6 (3.8) | -6.6 (3.0) | -6.0 (2.8) | -5.2 (4.1) | -6.0 (5.0) | -7.4 (4.3) | -6.9 (7.7) | -6.2 (3.7)
  Right hippocampus - Week 24 (n=4,6,6,5,5,6,8,6) | -7.3 (1.2) | -4.4 (4.7) | -6.3 (5.6) | -4.5 (7.1) | -5.1 (4.5) | -5.3 (2.4) | -6.5 (4.6) | -8.2 (5.0)

14. Secondary Outcome: Left and Right Hippocampal Cerebral Glucose Metabolism at Baseline and at Week 24
Description: Cerebral glucose metabolism was measured in validated 3 dimensional statistic surface projection analysis (Cortex ID®, GE Healthcare), transversal/coronal/sagittal-slice analysis (HERMES BRASS), and voxel-wise whole brain analysis (SPM5) using [18F]fluorodeoxyglucose positron emission tomography.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µCi/mL
Arm/Group | Placebo Every 2 Weeks | 0.1 g/kg Octagam 10% Every 2 Weeks | 0.25 g/kg Octagam 10% Every 2 Weeks | 0.4 g/kg Octagam 10% Every 2 Weeks | Placebo Every 4 Weeks | 0.2 g/kg Octagam 10% Every 4 Weeks | 0.5 g/kg Octagam 10% Every 4 Weeks | 0.8 g/kg Octagam 10% Every 4 Weeks
Number analyzed (Participants) | 7 | 6 | 6 | 6 | 6 | 7 | 8 | 7
µCi/mL
  Right hippocampus - Baseline | 0.83 (0.06) | 0.81 (0.06) | 0.81 (0.06) | 0.83 (0.06) | 0.81 (0.08) | 0.88 (0.03) | 0.82 (0.08) | 0.81 (0.04)
  Right hippocampus - Week 24 (n=6,6,6,5,3,6,8,6) | 0.84 (0.07) | 0.83 (0.07) | 0.83 (0.06) | 0.81 (0.02) | 0.82 (0.07) | 0.87 (0.04) | 0.84 (0.07) | 0.82 (0.03)
  Left hippocampus - Baseline | 0.79 (0.05) | 0.77 (0.06) | 0.80 (0.07) | 0.81 (0.05) | 0.81 (0.07) | 0.84 (0.05) | 0.80 (0.06) | 0.77 (0.04)
  Left hippocampus - Week 24 (n=6,6,6,5,3,6,8,6) | 0.80 (0.03) | 0.78 (0.05) | 0.84 (0.09) | 0.80 (0.07) | 0.81 (0.08) | 0.84 (0.05) | 0.81 (0.05) | 0.79 (0.05)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored throughout the entire study period, starting from the baseline visit until the final study visit.
Description: Safety set: All randomized participants who received at least 1 infusion of study medication.
Arm/Group | Placebo Every 2 Weeks | 0.1 g/kg Octagam 10% Every 2 Weeks | 0.25 g/kg Octagam 10% Every 2 Weeks | 0.4 g/kg Octagam 10% Every 2 Weeks | Placebo Every 4 Weeks | 0.2 g/kg Octagam 10% Every 4 Weeks | 0.5 g/kg Octagam 10% Every 4 Weeks | 0.8 g/kg Octagam 10% Every 4 Weeks
Serious Adverse Events (participants affected / at risk) | 2/7 | 1/6 | 0/7 | 2/7 | 2/7 | 0/7 | 1/8 | 0/7
Other Adverse Events (participants affected / at risk) | 5/7 | 4/6 | 5/7 | 3/7 | 3/7 | 4/7 | 4/8 | 4/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Every 2 Weeks (N=7) | 0.1 g/kg Octagam 10% Every 2 Weeks (N=6) | 0.25 g/kg Octagam 10% Every 2 Weeks (N=7) | 0.4 g/kg Octagam 10% Every 2 Weeks (N=7) | Placebo Every 4 Weeks (N=7) | 0.2 g/kg Octagam 10% Every 4 Weeks (N=7) | 0.5 g/kg Octagam 10% Every 4 Weeks (N=8) | 0.8 g/kg Octagam 10% Every 4 Weeks (N=7)
Gastral antral vascular ectasia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Knee arthroplasty (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal laminectomy (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dementia Alzheimer's Type (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aggression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Every 2 Weeks (N=7) | 0.1 g/kg Octagam 10% Every 2 Weeks (N=6) | 0.25 g/kg Octagam 10% Every 2 Weeks (N=7) | 0.4 g/kg Octagam 10% Every 2 Weeks (N=7) | Placebo Every 4 Weeks (N=7) | 0.2 g/kg Octagam 10% Every 4 Weeks (N=7) | 0.5 g/kg Octagam 10% Every 4 Weeks (N=8) | 0.8 g/kg Octagam 10% Every 4 Weeks (N=7)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Iron deficiency anemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colitis microscopic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Submandibular mass (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anxiety postoperative (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Post procedural constipation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Procedural headache (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Procedural hypertension (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood iron decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood pressure decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
CSF white blood cell count positive (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Essential tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Hypertonia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hyporeflexia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood pressure fluctuation (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vasoconstriction (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Small numbers of patients per treatment group (between 5 and 8) and variable total Aβ levels over time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No